CLINICAL TRIAL: NCT01455571
Title: Phase I Study to Determine the Maximum Tolerated Dose and to Assess the Safety and Pharmacokinetic Profile of HM781-36B
Brief Title: Phase I Study to Determine the Maximum Tolerated Dose and to Assess the Safety and Pharmacokinetic Profile of HM781-36B in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Collaborators: Seoul National University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-PHI-101
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM781-36B (Experimental): Dose : 0.5mg, 1mg, 2mg, 4mg, 8mg, 12mg, 16mg, 20mg,...
  Interventions: Drug: HM781-36B

INTERVENTIONS:
Drug: HM781-36B — Q1DX14/2W for 3W HM781-36B

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) of HM781-36B.

DETAILED DESCRIPTION:
Besides the main objective, there are 3 other objectives as follows:

1. To determine dose-limiting toxicity (DLT) of HM781-36B
2. To characterize the pharmacokinetics of HM781-36B, following oral administration of HM781-36B
3. To evaluate anticancer activity of HM781-36B in patients with advanced solid malignancies Groups of 3 patients per cohort or dose level will be treated with escalating doses of HM781-36B

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologically or cytologically confirmed advanced solid tumor 2) Patients who have experienced progressive disease despite of conventional anticancer therapy. Patients who cannot expect effective treatment or prolonged survival with conventional anticancer therapy 3) Previous chemotherapy, radiotherapy and surgical operation are allowed if they are discontinued for at least 4 weeks prior to D0 and all adverse events are resolved 4) Aged ≥19 5) Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2 6) A life expectancy greater than 12 weeks 7) Adequate bone marrow (WBC≥4,000/mm3 platelet≥100000/mm3, hemoglobin≥9.0g/dl and ANC≥ 1500/mm3, renal (Creatinine≤1.5mg/dl) and liver function (AST/ALT/ALP ≤ 3 x upper limit of normal and total bilirubin≤2mg/dl) and no abnormal heart and lung function However, AST/ALT/ALP ≤ 5 x upper limit of normal for patients with liver metastases and ALP level ≤ 5 x upper limit of normal for patients with bone metastases are allowed 8)Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

* 1) Patients with hematopoietic malignancies,uncontrolled infection, ileus, CNS metastasis.

  2) Patients who have undergone hematopoietic stem cell transplantation (HSCT) or are candidates for planned HSCT 3) Class III or IV heart failure (NYHA Class) or LVEF<40% 4) Patients who have GI malabsorption or difficulty taking oral medication 5) Patients who have psychiatric or congenital disorder 6) Subjects who, in the investigator's opinion, cannot be treated per protocol due to functional impairments 7) Pregnant or breast-feeding patients; Women of childbearing potential without adequate contraception (Men must use adequate contraception.) 8) Subjects who have no intention of following the requirements of the protocol or the follow-up management. Subjects who cannot be followed up regularly due to psychological, social, family, logistic, and geographical reasons 9) Subjects who were administered with other investigational products within 30 days before screening.

  10) Subjects who, in the investigator's opinion, cannot be participated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
MTD determination | Dose limiting Toxicity will be evaluated on Day 21 during Cycle 1

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea